CLINICAL TRIAL: NCT00887705
Title: Activities of Daily Living (ADL)-Training for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ADL- Training for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LHL Helse (Other)
Responsible Party: Morten Ryg, Glittreklinikken
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GK-63
Record Dates: First submitted 2009-04-14; First posted 2009-04-24 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary Rehabilitation; ADL-Training; COPD Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Standard rehabilitation programme (No Intervention)
- 2. Additional ADL training (Experimental)
  Interventions: Behavioral: ADL training

INTERVENTIONS:
Behavioral: ADL training — The control group gets the standard rehabilitation programme which includes one hour ADL- training. The experimental group also gets the standard rehabilitation program, but instead of one hour they get an additional five hours ADL- training.
  Arms: 2. Additional ADL training

SUMMARY:
ADL training of copd patients results in better execution of activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Referred for rehabilitation
* Age > 18 years
* Symptoms affecting ADL function
* 6 minute walk distance (6MWD) < 400 meters

Exclusion Criteria:

* Patients who smokes or has smoked during the last three months.
* LTOT
* Patients who has another disability
* Patients who can't read or speak Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure(COPM) - Self-perception of occupational performance and satisfaction. | Baseline, 4 weeks; 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Morten S Ryg, Dr philos, Study Director — LHL Helse
Locations (2):
- Norway (2):
  - Glittreklinikken, Hakadal, Akershus
  - Glittreklinikken, Hakadal

REFERENCES:
- See also: Site of LHL (Norwegian association for lung and heart disease patients). Glittreklinikken is listed as part of the organization — http://www.lhl.no